### Official Title of Study:

An Investigational Study of Continuous 8-Hour Intravenous Administrations of BMS-986231 in Participants With Heart Failure and Reduced Heart Function Given a Standard Dose of Loop Diuretic

NCT Number: NCT03730961

Document Date (Date in which document was last revised): January 22, 2020

Version Date: 22-Jan-2020

## **Statistical Analysis Plan**

| Sponsor: | Bristol-Myers Squibb Research and Development |
|---|---|
| Protocol No: | CV013-034 |
| Protocol Title: | A Randomized, Double-Blind, Placebo-Controlled, Cross-over Phase 2<br>Study of Continuous 8-Hour Intravenous Infusions of BMS-986231 in<br>Patients with Heart Failure and Impaired Systolic Function Given a<br>Standard Dose of Loop Diuretic |
| PRA Project ID: | BMS001PC-180016 |

### 1.0 Approvals

The undersigned have approved this Statistical Analysis Plan for use in this study.



EDSREP 009 T 01 G 





### 2.0 Table of Contents

| 1.0 Approvals | |
|-------------------------------------------------------|------|
| 2.0 Table of Contents | |
| 3.0 Introduction | 4 |
| 4.0 Changes from Previous Version of Approved SAP | 4 |
| 5.0 Study Objectives | 4 |
| 5.1 Primary | 4 |
| 5.1.1 Primary Endpoints | 4 |
| 5.2 Secondary | 4 |
| 5.2.1 Secondary Endpoints | |
| 5.2.2 Safety Endpoint | 4 |
| 3.0 Study Design | |
| 6.1 Sample Size Considerations | |
| 6.2 Randomization | |
| 7.0 Overview of Planned Analysis | 6 |
| 7.1 Changes from Protocol | 6 |
| 7.2 Planned Analyses | |
| 7.2.1 Preliminary Analysis | 6 |
| 7.2.2 Topline Results | |
| 7.2.3 Final Analysis | |
| B.0 Definitions and General Analysis Methods | 7 |
| 8.1 Analysis Data Presentation | |
| 8.1.1 Rounding | 7 |
| 8.1.2 Imputation | |
| 8.1.3 Descriptive Statistics | 7 |
| 8.1.4 Pooling | 7 |
| 8.1.5 Unscheduled Measurements | 7 |
| 8.2 Analysis Data Definitions | 8 |
| 8.2.1 Baseline Definition | |
| 8.2.2 Treatment/Subject Grouping | |
| 8.2.3 Common Variable Derivations | |
| 8.2.4 QC | |
| 8.2.5 ADaM Datasets and Metadata | 8 |
| 8.3 Software | |
| 8.4 Statistical Methods | |
| 8.4.1 Statistical Outlier Determination | |
| 8.4.2 Predetermined Covariates and Prognostic Factors | |
| 8.4.3 Hypothesis Testing | 9 |
| 9.0 Analysis Sets | 6 |
| 9.1 Enrolled | |
| 9.2 Randomized | |
| 9.3 Treated (per protocol) | |
| 9.4 Safety | |
| 10.0 Subject Disposition | |
| 11.0 Protocol Deviations | |
| 12.0 Demographic and Baseline Characteristics | |
| 12.1 Demographics | |
| 12.2 Medical History | |
| • | . 10 |
| 14.0 Treatment Compliance and Exposure | . 10 |
| 15.0 Efficacy Analyses | |





| 15.1 Effect of BMS-986231 on urine output | |
|---|---|
| 15.2 Effect of BMS-986231 on fractional excretion | 11 |
| 15.3 Effect of BMS-986231 on furosemide concentration | 11 |
| 16.0 Pharmacokinetic Analyses | 12 |
| 16.1.1 Plasma Concentrations | 12 |
| 16.1.2 Urine Concentrations | 12 |
| Safety Analyses | 13 |
| 16.2 Safety Variables | 13 |
| 16.2.1 Adverse Events | |
| 16.2.2 Deaths and Serious Adverse Events | |
| 16.2.3 Laboratory Data | 14 |
| 16.2.4 Vital Signs | |
| 16.2.5 Electrocardiograms | 14 |
| 16.2.6 Physical Examinations | 14 |
| Appendix 1: Glossary of Abbreviations | 16 |
| Appendix 2: Schedule of Activities from Protocol | 17 |
| Appendix 3: Blood Sampling and Urine Collection Intervals for PK and Efficacy | |
| Appendix 4: List of Tables, Figures, and Listings | |
| Appendix 6: Shells for Tables, Figures and Listings | 28 |
| 18.0 Document History | 29 |


### 3.0 Introduction

This Statistical Analysis Plan (SAP) describes the statistical methods that will be used during the analysis and reporting of data collected under Bristol-Myers Squibb Research and Development (BMS) Protocol CV013034.

This SAP should be read in conjunction with the study protocol and electronic case report form (eCRF). This version of the plan has been developed using the protocol dated 15-Apr-2019 (including all amendments up to this date) and the final eCRF(s) dated 22-Oct-2018.

An approved and signed SAP is a requirement for database lock.

This SAP only covers the results that will be processed by the PRA Early Development Services (EDS) Biostatistics Department.

PRA EDS will perform the efficacy, pharmacokinetic (PK), pharmacodynamic (PD), biomarker and safety and tolerability evaluations.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. Any post-hoc or unplanned analyses, or significant changes from the planned analysis in this SAP performed to provide results for inclusion in the clinical study report (CSR) but not included in this SAP, will be clearly identified in the CSR. Changes to planned analyses do not require an updated SAP but should be discussed with the sponsor and included in the CSR if significant.

### 4.0 Changes from Previous Version of Approved SAP

This is the first version of the SAP.

### 5.0 Study Objectives

### 5.1 Primary

Evaluate the effects of HNO donor BMS-986231 on 4-hour urine output in patients with HFrEF after administration of 40 mg of IV furosemide.

### 5.1.1 Primary Endpoints

The total volume of urinary output 4 hours after 40 mg furosemide bolus given to patients with HFrEF while on BMS-986231 compared to placebo: absolute difference in total volume and % change from placebo.

### 5.2 Secondary

Assess the effect of BMS-986231 on fractional excretion of Na (FeNa)

Assess the effect of BMS-986231 on fractional excretion of K (FeK)

Assess the effects of BMS-986231 on furosemide urinary and plasma concentration and the ratio urinary sodium to urinary furosemide

Assess safety of BMS-986231

### 5.2.1 Secondary Endpoints

FeNa, FeK, furosemide urinary and plasma concentration and ratio urinary sodium to urinary furosemide at 8 hours post-start infusion. Parameter values while patient is on BMS-986231 compared to placebo: absolute differences and % change from placebo.

### 5.2.2 Safety Endpoint

Clinically relevant hypotension (defined as SBP < 90 mmHg or symptomatic hypotension) during infusion, incidence of AEs, abnormal clinical laboratory values, vital signs, ECGs, telemetry, physical examinations.

EDSREP 009 T 01 G 



Protocol: CV013-034



### 6.0 Study Design

This is a double blinded, randomized, two-way cross-over, placebo-controlled study to evaluate the effects of HNO donor BMS-986231 on 4-hour urine output in HFrEF patients after administration of 40 mg of IV furosemide. The study consists of 2 one-day treatment periods (BMS-986231 or placebo) separated by a washout period of at least 7 days (Day 2 to at least Day 8), but no more than 4 weeks. Each period includes 8-hour infusion. A standard dose of 40 mg IV furosemide will be administered by IV bolus injection at the midpoint (4 hour, H4) of an 8-hour infusion. Screening for inclusion in the study will be performed up to 4 weeks before the first treatment day (Day 1 of the first period). Approximately 20 subjects will be included. The total duration of the study will be approximately 8 weeks.

### **Study Design Schematic from Protocol:**

EDSREP 009 T 01 G 







### 6.1 Sample Size Considerations

The number of subjects to be enrolled was chosen based on practical considerations. Twenty patients with HFrEF will be randomized to one of 2 sequences: BMS-986231/furosemide followed by placebo/furosemide or placebo/furosemide followed by BMS-986231/furosemide. The difference between BMS-986231 and placebo in total urine output in the 4 hours following furosemide administration will be estimated and presented with 95% confidence intervals (CIs).

Normal healthy volunteers have a urinary output around 0.5-1.0 mL/kg/H (40-100 mL/H), which could be decreased in people over 65 years old or patients with HF at around 0.2-0.5 mL/kg/H (20-40 mL/H). Patients with HF given a bolus of IV loop diuretics is estimated to have their diuresis increased to 250-300 mL/H in the 4 hours following the administration. Assuming the standard deviation of urine output change is 20~35 mL/H based on the estimated range of the changes, with 20 patients, the study will be able to demonstrate a 20% increase in urinary output compared to placebo, with 90% power.

### 6.2 Randomization

The subjects were randomized by the Biostatistics Department of the EDS group of PRA Health Sciences using PROC PLAN in SAS. Subjects (N=20 plus 4 additional) were assigned to one of the two sequences active treatment/placebo or placebo/active treatment with a 1:1 allocation ratio. An additional randomization was run a second time for the second site (Richmond, London) which was only added to the study when it was already running at the first site (NHS, Glasgow). For details, please see Global Note to File no.2.

Subject numbers that were used are R01-R24 and S01-S24. Participants will not be replaced if they are discontinued from the study.

### 7.0 Overview of Planned Analysis

### 7.1 Changes from Protocol

There are no changes from protocol

### 7.2 Planned Analyses

### 7.2.1 Preliminary Analysis

No preliminary analysis is planned.

EDSREP 009 T 01 G 


### 7.2.2 Topline Results

Topline tables, figures, and listings (TFLs) will be provided after database lock. Topline TFLs will be determined by the Biostatistics Asset Lead and Clinical Pharmacology Asset Lead prior to programming commencing and will be the minimal set of TFLs needed to analyze key endpoints.

### 7.2.3 Final Analysis

The full set of draft TFLs will be provided after topline TFLs. After comments have been incorporated on the draft TFLs, the TFLs will be approved by the Biostatistics Asset Lead and incorporated in the CSR.

### 8.0 Definitions and General Analysis Methods

### 8.1 Analysis Data Presentation

### 8.1.1 Rounding

In listings, data will be presented with the same precision as the original data. Derived data will be rounded for presentation purposes.

For all summaries (with the exception of PK), the mean will be presented to 1 decimal greater than the original data, the SD to 2 decimals greater than the original data, and the median, minimum (min) and maximum (max) values will be presented to the same number of decimal places as the original data.

For PK summaries, mean, SD, median, min, and max values  $\geq$  100 will be presented as integers, values < 100 but  $\geq$  10 will be presented with 1 decimal, values < 10 but  $\geq$  1 will be presented with 2 decimals, and values < 1 will be presented with 3 decimals. Ratios will be presented with 3 decimals. Coefficient of variation (%CV) will be presented with 1 decimal.

For listing presentation purposes, PK parameters will be rounded in the same manner as noted above for summaries.

P-values will be reported to 4 decimal places; p-values less than 0.0001 will be reported as p <0.0001.

### 8.1.2 Imputation

Unless otherwise noted, data will not be imputed.

### 8.1.3 Descriptive Statistics

Unless otherwise indicated in specific data type sections, continuous variables will be summarized with the following descriptive statistics: n (number of observations), (arithmetic) mean, SD, median, min, and max.

Categorical data will be summarized with frequencies and percentages. Percentages by categories will be based on the number of subjects within a treatment group. Percentages will be rounded to 1 decimal, except 100% which will be displayed without any decimal places. Percentages will not be displayed for zero counts. Categories will be presented in the tables exactly as they appear in the CRF / Database.

### 8.1.4 Pooling

No data will be pooled for this study.

### 8.1.5 Unscheduled Measurements

Unscheduled measurements will be included in the listings. With the exception of unscheduled measurements used for baseline, unscheduled measurements will be excluded from the descriptive statistics and statistical analysis.

EDSREP 009 T 01 G 


### 8.2 Analysis Data Definitions

### 8.2.1 Baseline Definition

Unless otherwise stated, baseline for post-dose evaluations is defined as the last observation recorded before the study drug administration in a period. The last observation can be an unscheduled / repeated measurement.

### 8.2.2 Treatment/Subject Grouping

| Label | Grouping |
|---|---|
| Study Drug | BMS-986231 or Placebo |
| Treatment | BMS-986231: BMS-986231 12 $\mu g/kg/min$ for 8 hours (20 mL/H), single infusion IV |
| | Placebo: Placebo 20 mL/H for 8 hours, single infusion IV |
| | Furosemide: Furosemide 40 mg, single IV bolus |

### 8.2.3 Common Variable Derivations

| Variable | Dataset | Definition/Calculation |
|---|---|---|
| Change from Baseline | All | Post-dose Observation minus Baseline Observation |
| Analysis Period | All | Interval of time during which treatment is constant. |
| TEAE | AE | AE is a TEAE if the AE Date/Time is greater than or equal to the first Dose Date/Time |

### 8.2.4 QC

The analysis datasets and the TFLs will be QC'd according to the PRA EDS QC plan that is developed according to the EDSREP 009 SOP.

### 8.2.4.1 Critical Data

The QC plan requires datasets be classified as critical or non-critical. The datasets considered critical are subject level, efficacy, and adverse events (ADSL, ADEFF, and ADAE).

### 8.2.5 ADaM Datasets and Metadata

The analysis datasets will be generated in accordance with Clinical Data Interchange Standard Consortium (CDISC) Analysis Data Model (ADaM) Version 2.1.

ADaM compliant datasets will be delivered to the sponsor. A define.xml file version 2 with the corresponding metadata will be included. Analysis results metadata are excluded.

### 8.3 Software

The statistical analysis and reporting will be done using SAS<sup>®</sup> for Windows<sup>™</sup> Version 9.4 or higher (SAS Institute, Inc.).

PK parameter calculations will primarily be done using Phoenix<sup>®</sup> WinNonlin<sup>®</sup> Version 8.1 or higher (Certara, Inc.). Additional PK computations may be performed in SAS<sup>®</sup>.

EDSREP 009 T 01 G 


### 8.4 Statistical Methods

### 8.4.1 Statistical Outlier Determination

No statistical outlier analysis is planned.

### 8.4.2 Predetermined Covariates and Prognostic Factors

There are no predetermined covariates or prognostic factors.

### 8.4.3 Hypothesis Testing

Unless otherwise stated, all significance testing will be 2-sided at the significance level of 0.05.

### 9.0 Analysis Sets

| Analyses | Enrolled | Randomized | Treated per protocol | Safety |
|---|---|---|---|---|
| Disposition | ✓ | | | |
| Baseline<br>Characteristics | | ✓ | ✓ | |
| Safety Assessments | | | | ✓ |
| Primary Efficacy<br>Analysis | | | ✓ | |
| Other Efficacy<br>Analysis | | | ✓ | |
| PK Analysis | | | ✓ | |

### 9.1 Enrolled

All participants who sign informed consent.

### 9.2 Randomized

All randomized subjects who have started study drug infusion in at least one treatment period. This is also known as the Intent to Treat (ITT) population. Data in this data set will be analyzed based on randomized sequence of treatments.

### 9.3 Treated (per protocol)

All randomized participants who were given both study treatments and completed the study as per protocol. Participants will be included in the treatment group they received in each period.

### 9.4 Safety

All randomized participants who take at least 1 dose of double-blind study treatment. Participants will be included in the treatment group they received in each period.

### 10.0 Subject Disposition

The number of subjects in each analysis set will be presented.

The number and percentage of subjects who withdrew from the study prematurely and a breakdown of the corresponding reasons for withdrawal will be presented by analysis set. Percentages will be based on the total number of subjects in the analysis set.

EDSREP 009 T 01 G 


### 11.0 Protocol Deviations

Protocol deviations will be collected and entered into the Clinical Trial Management System (CTMS) per clinical monitoring Standard Operating Procedures. From CTMS, protocol deviations will be pulled into SDTM. Important protocol deviation data will be listed by subject.

### 12.0 Demographic and Baseline Characteristics

### 12.1 Demographics

Subject demographics will be summarized descriptively for the Randomized and Per Protocol analysis sets. The summary will include the subjects' age (years), sex, race, ethnicity, weight (kg), height (cm), and BMI (kg/m²). Any measurements will be included from assessments performed during the Screening Visit.

All demographic data, as collected during the screening visit, will be listed by subject.

### 12.2 Medical History

Medical history including disease under study will be categorized by preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) and will be listed by subject.

### 12.3 Other Baseline Characteristics

All screening criteria data collected on the CRF (including failed eligibility criteria) will be listed by subject. Childbearing Potential will be listed.



### 14.0 Treatment Compliance and Exposure

The number and percentage of subjects receiving full dose of study drug will be summarized by sequence in periods 1 and 2 for the safety analysis set.

All study drug administration data will be listed by subject.

### 15.0 Efficacy Analyses

### 15.1 Effect of BMS-986231 on urine output

All primary efficacy analyses will be performed using the treated (per protocol) population.

Urinary output will be listed by timepoint.

The volumes (total within 4 h after furosemide dosing, total within 4 h before furosemide dosing, total within 8 h after start of BMS-986231/placebo dosing and difference of totals after and before furosemide dosing) after BMS-986231 and after placebo will be calculated per patient.

Descriptive statistics (n, mean, SD, %CV, median, min, and max) will be used to summarize the absolute difference between the volumes under BMS-986231 dosing and under placebo and the percent change from placebo under BMS-986231 dosing of urinary output by treatment.

EDSREP 009 T 01 G 


Plots of the arithmetic mean urinary output + SD by scheduled sampling times will be provided by treatment. Bar plots showing the arithmetic mean urinary output and the individual urinary output by interval and treatment will be provided. These plots will show time in hours. The plots will match the summary table results. Plots will be presented to the last scheduled time point.

A within patient analysis using a paired T-test will be performed to compare the volumes of urinary excretion and to test if there is a significantly different amount of urine secreted while receiving BMS-986231 versus placebo. Body weight might be considered as covariate, if significant.

### The SAS PROC TTEST code is as follows:

```
proc ttest data = volume;
    PAIRED BMS-986231*placebo;
run;
```

Paired profiles and Q-Q plot of the urinary output under BMS-986231 and placebo treatment will be provided for a visual representation of the data.

### 15.2 Effect of BMS-986231 on fractional excretion

Secondary efficacy analyses will be performed using the per protocol population.

The fractional excretion (total within 4 h after furosemide dosing, total within 4 h before furosemide dosing, total within 8 h after start of BMS-986231/placebo dosing and difference of totals after and before furosemide dosing) of Na (FeNa) and K (FeK) after BMS-986231 and after placebo will be calculated per patient.

Descriptive statistics (n, mean, SD, %CV, median, min, and max) will be used to summarize the absolute difference between the excretion under BMS-986231 dosing and under placebo and the percent change from placebo under BMS-986231 dosing of fractional excretion by treatment.

Bar plots showing the arithmetic mean urinary output and the individual urinary output by interval and treatment will be provided.

A within patient analysis using a paired T-test will be performed to compare the volumes of urinary excretion and to test if there is a significantly different amount of urine secreted while receiving BMS-986231 versus placebo.

Paired profiles of fractional excretion will be provided for a visual representation of the data.

### 15.3 Effect of BMS-986231 on furosemide concentration

Furosemide urinary and plasma concentrations and the ratio of urinary sodium to urinary furosemide will be calculated at each time point over 4-hour urine/plasma collection after a bolus injection of 40 mg furosemide while receiving BMS-986231 or placebo

Descriptive statistics (n, mean, SD, %CV, median, min, and max) will be used to summarize the absolute difference and the percent change from placebo of furosemide urine concentration, furosemide plasma concentration and the ratio of urinary sodium to urinary furosemide at 8 h by treatment.

Paired profiles of furosemide urine concentration, furosemide plasma concentration and the ratio of urinary sodium to urinary furosemide (4 h after furosemide dosing) will be provided for a visual representation of the data.



EDSREP 009 T 01 G 



Protocol: CV013-034



### 16.0 Pharmacokinetic Analyses

The PK summaries described in this section will be created using the Randomized analysis set.

### **16.1.1 Plasma Concentrations**

Descriptive statistics (n, mean, SD, CV%, geometric mean, median, min, and max) will be used to summarize the plasma concentrations of Furosemide, BMS-986231 (and its metabolites) at each scheduled time point (see table in Appendix 3).

Plasma concentrations below the limit of quantification (BLQ) will be set to missing in the computation of mean concentration values. No descriptive statistics will be provided if more than half of the subjects have values BLQ.

All individual subject plasma concentration data will be listed.

### **16.1.2 Urine Concentrations**

Urine recovery of Furosemide, BMS-986231 (and its metabolites) will be calculated per interval and cumulative. Parameters will be calculated as follows for 4-10 h for furosemide and for 0-10 h for BMS-986231 and metabolites:

| Parameter | Description | SAS Programming<br>Notes |
|---|---|---|
| Ae(0-T) | Cumulative amount of drug excreted unchanged into urine to time t (last scheduled sample). | Summation i = 1 to n of (Concentration |
| | The amounts recovered in urine over a collection interval are calculated by multiplying the urine concentrations for each analyte by the total volume/weight of the sample collected during that interval. | (ng/mL) t <sub>i-1</sub> -<br>t <sub>i</sub> *volume(mL)t <sub>i-1</sub> -t <sub>i</sub> ) |
| | The sum of the amount recovered for all intervals is calculated to obtain the total amount recovered in urine, obtained by adding the amounts excreted over each collection interval. | |

EDSREP 009 T 01 G 


| Parameter | Description | SAS Programming<br>Notes |
|---|---|---|
| Fe | Fraction (represented in %) of the administered dose excreted unchanged into urine. The sum of the percentage of dose for each analyte for all intervals will be calculated to obtain the total percentage urinary recovery. | (Ae(0-T)/Dose)*100 |

All individual subject urine parameters (interval times, concentration, volume, amount excreted in interval) data will be listed.

Otherwise urine parameters will be summarized as described above.

### **Safety Analyses**

The safety summaries described in this section will be created using the Safety set.

### 16.2 Safety Variables

The following safety variables will be included:

- Adverse Events
- Clinical Laboratory Evaluations
- Vital Signs
- Electrocardiograms

### 16.2.1 Adverse Events

An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant that does not necessarily have a causal relationship with treatment. Treatment-emergent adverse events (TEAEs) are those which occur after the first dose of study drug. All TEAE summaries will be presented alphabetically by system organ class, with preferred terms sorted in decreasing order of frequency within each system organ class based on MedDRA dictionary.

For treatment period assignment, the following rules will be applied:

- TEAEs occurring following dosing in period 1 but before dosing in period 2 will be attributed to the drug administered in period 1.
- TEAEs occurring following dosing in period 2 will be attributed to the drug administered in period 2

If the time is missing for an AE on a dosing day, then the AE will be attributed to the treatment period of the treatment given on that day.

The following missing data will be imputed (for calculations only) as defined:

- Missing AE start and / or end times for the calculation of onset and duration will be assumed to be at 00:01 for a start time and 23:59 for end times
- Missing AE severity or relationship will be left as missing
- Missing AE start times for the determination of treatment emergence will be assumed to occur after treatment unless partial date documents the AE as happening prior to treatment
- Missing AE start times for the determination of treatment assignment will be assumed to occur after treatment on the recorded date one minute after dosing
- Missing AE start date will be assumed to be after treatment for the determination of TEAE but will
  not be attributed to a specific treatment

EDSREP 009 T 01 G 


A summary of the number and percentage of subjects reporting AEs, TEAEs by severity, serious AEs (SAEs), and who discontinue study drug due to an AE will be presented by treatment and overall.

A summary of the number and percentage of subjects reporting each TEAE will be presented by treatment and overall. Counting will be done by subject only, not by event; subjects will only be counted once within each body system or preferred term.

A summary of the number and percentage of subjects reporting each TEAE will be presented by relationship to BMS-986231 (as recorded on the CRF) and by treatment and overall. Subjects with multiple events will be counted under the category of their most-related event within each system organ class or preferred term.

A summary of the number and percentage of subjects reporting each TEAE will be presented by relationship to Furosemide (as recorded on the CRF) and by treatment and overall. Subjects with multiple events will be counted under the category of their most-related event within each system organ class or preferred term.

A summary of the number and percentage of subjects reporting each TEAE will be presented by severity (as recorded on CRF) and by treatment and overall. Subjects with multiple events will be counted under the category of their most severe event within each system organ class or preferred term.

All AEs (including non-treatment-emergent events) recorded on the eCRF will be listed by subject.

A separate listing of AEs leading to study drug discontinuation will be provided by subject.

### 16.2.2 Deaths and Serious Adverse Events

A listing of deaths and other SAEs will be provided by subject.

### 16.2.3 Laboratory Data

Clinical laboratory data will be presented using Système International (SI) units from the study data tabulation model (SDTM) Controlled Terminology.

A descriptive statistics summary of continuous laboratory results for chemistry and hematology and derived changes from baseline will be provided by scheduled time point.

All laboratory data will be listed by subject, including laboratory variables not listed in the protocol.

A separate listing of out-of-range values will also be provided. Normal ranges will be used directly from the clinical laboratory and will be included in the listings for reference.

Results from pregnancy tests will be listed.

### 16.2.4 Vital Signs

A descriptive statistics summary of vital signs and derived changes from baseline will be provided by treatment and scheduled time point.

All vital signs data will be listed by subject. A separate listing of hypotension will be provided.

### 16.2.5 Electrocardiograms

The observed measurements for all ECG parameters and the corresponding abnormalities will be listed for all timepoints. The means of triplicate measurements for continuous parameters and the change from baseline of the mean triplicate measurements at each scheduled timepoint will be listed by subject.

Descriptive statistics will be provided to summarize mean ECG parameters (observed and changes from baseline) by treatment and scheduled time.

### 16.2.6 Physical Examinations

All physical examination data will be listed by subject.

EDSREP 009 T 01 G 


EDSREP 009 T 01 G 




### **Appendix 1: Glossary of Abbreviations**

| Glossary of Abbreviation | ns: |
|--------------------------|-----------------------------------------------|
| AE | Adverse event |
| ADaM | Analysis data model |
| BLQ | Below the limit of quantification |
| BMI | Body mass index |
| BMS | Bristol-Myers Squibb |
| CDISC | Clinical Data Interchange Standard Consortium |
| CI | Confidence interval |
| CSR | Clinical study report |
| CTMS | Clinical Trial Management System |
| CV | Coefficient of variation |
| DDT | Data definition table |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EDS | Early Development Services |
| LLOQ | Lower limit of quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| SAP | Statistical analysis plan |
| SAE | Serious adverse event |
| SDTM | Study data tabulation model |
| TEAE | Treatment-emergent adverse event |
| TFL(s) | Tables, figures and listings |
| WHO | World Health Organization |

EDSREP 009 T 01 G 

Protocol: CV013-034 Version Date: 22-Jan-2020



Appendix 2: Schedule of Activities from Protocol

Table 1: Screening Procedural Outline (CV013-034)

| | Scroonin | |
|---|---|---|
| Procedure | g<br>Visit | Notes |
| Eligibility Assessments | | |
| Informed Consent | × | A participant is considered enrolled only when a protocol specific informed consent is signed. |
| Inclusion/Exclusion Criteria | × | |
| Medical History | × | |
| Safety Assessments | | |
| Physical Examination | × | If the screening physical examination is performed within 3 days prior to first dosing then a single exam may count as both the screening and predose evaluation. Includes height, and BMI. |
| Vital Signs | × | Includes body temperature, respiratory rate, and seated blood pressure and heart rate. Blood pressure and heart rate should be measured after the participant has been resting quietly for at least 5 minutes. |
| Adverse Events Assessment | × | SAEs must be collected from the date of the participant's Informed consent. |
| ECG | × | ECGs should be recorded after the participant has been supine for at least 5 minutes. At screening, single ECGs will be recorded. |
| Laboratory Tests | × | Includes blood (hematology, serum chemistry, NT-proBNP or BNP [details in the protocol section]) and urine samples. Participants are required to fast for at least 10 hours prior to the collection of specimens for clinical laboratory tests (details in the protocol Section 8.4.6). |
| Pregnancy Test | × | For |

 EDSREP 009 T 01 G BMS001PC-180016 Protocol: CV013-034 Version Date: 22-Jan-2020

# Table 2: On Treatment Procedural Outline (CV013-034)

| | L | Treatment Period | ро | Notes |
|---|---|---|---|---|
| Procedure | Period 1<br>Day 1 | Washout<br>(7-28 days) | Period 2<br>Day 1 | Washout between periods should be at least 7 days and no more than 4 weeks. |
| Safety Assessments | | | | |
| Weight | × | | × | Weight within 15 minutes prior to and within 15 minutes after the end of the infusion in each treatment period with bio-impedance scale. Weight should be measured after the void. |
| Targeted physical examination | × | | × | To be done at H0 (before start of infusion). Based on subject's report since the last visit. Includes temperature, signs and symptoms of congestion. If the screening physical examination is performed within 3 days prior to first dosing then a single physical exam may count as both the screening and at H0 (before start of infusion) evaluation. |
| Vital Signs<br>(Blood pressure and heart rate) | × | | × | Prior to infusion, and 30 minutes for first hour then every 1 hour until discontinuation of infusion, then at H9, H10 and H11.5 (3.5 hour after end of infusion) in each treatment period. |
| Peripheral Oxygen Saturation | × | | × | Prior to the start of infusion and immediately prior to the end of the infusion in each treatment period, measured with a pulse oximeter device. |
| 12-lead ECG | × | | × | Prior to the infusion and after end of infusion (both with 15 minutes window) in each treatment period. Triplicate ECGs will be recorded. |
| Telemetry | × | | × | From start of infusion to 3 hours after end of infusion in each treatment period. |
| Adverse Events Assessment | × | | × | Nonserious AEs will be collected from the start of the study drug infusion until 24 hours after end of infusion in each treatment period of dosing. Serious adverse events must be collected from the date of Informed consent and will be assessed up to 30 days after end of infusion of the last period. |
| | | - | - | |
| Follow-up call/assessment | × | | × | To be done at Day 2 of each period. Will inquire about general status and occurrence of any AEs. |

 EDSREP 009 T 01 G



BMS001PC-180016 Protocol: CV013-034 Version Date: 22-Jan-2020

# On Treatment Procedural Outline (CV013-034)

Table 2:

| | | Treatment Period | ро | Notes |
|---|---|---|---|---|
| Procedure | Period 1<br>Day 1 | Washout<br>(7-28 days) | Period 2<br>Day 1 | Washout between periods should be at least 7 days and no more than 4 weeks. |
| | | | | For each period, subjects must remain for at least 3.5 hours after the end of infusion. Patients may stay overnight or may be discharged the same day 3.5 hours after end of infusion if certain conditions are met |
| Laboratory Tests | | | | |
| Hematology and Serum<br>Chemistry | × | | × | Laboratory tests will be performed in the morning of each treatment day (H0 [before start of infusion], H4 [just before furosemide bolus], and H8). |
| Pregnancy Test (WOCBP only) | × | | × | |
| Blood sampling for PK<br>(furosemide and BMS-986231<br>[and its metabolites]) | × | | × | Blood sampling for PK will be done at H0 (before start of infusion), H2 and at H4 hours (just before furosemide bolus), H5, H6, H8 (or end of infusion) and H10 (2 hours after the end of the infusion) in each treatment period. In addition, PK samples should be taken when the dose is lowered or discontinued |
| Blood sampling for Na, K, bicarbonate, creatinine, and eGFR | × | | × | Blood sampling for Na, K, bicarbonate, creatinine, and eGFR will be done at H0 (before start of infusion), H4 (just before furosemide bolus), H5, H6, H7, H8 (or end of infusion) in each treatment period. |
| Urine sampling for furosemide and BMS-986231 (or its metabolites) | × | | × | Urine samples can be taken from the urine collection intervals done for the urinary output. An aliquot for both sets of metabolites and a back-up will be required for the analysis. |
| Urine sampling for Na, K, P, CI, creatinine and bicarbonate concentrations | × | | × | Urine samples can be taken from the urine collection intervals done for the urinary output. |
| Efficacy Assessments | | | | |
| Urinary output | × | | × | Prior to start of infusion, patients will be asked to void and urine collected. A bladder scan (ultrasound) could be performed to ensure adequate bladder emptying. Patients will be asked to void at least every 2 hours during the first 4 hours post-start infusion and before furosemide bolus, and at least hourly from 4 to 8 hours post-start infusion. A second bladder scan could be performed at H8 (8 hours after start of infusion and just after study drug discontinuation and after the void). |

 EDSREP 009 T 01 G Protocol: CV013-034 Version Date: 22-Jan-2020



On Treatment Procedural Outline (CV013-034)

Table 2:

| - | F | Treatment Period | ро | Notes |
|---|---|---|---|---|
| Procedure | Period 1 | Washout | Period 2 | Washout between periods should be at least 7 days |
| | Day 1 | (7-28 days) | Day 1 | and no more than 4 weeks. |
| | | | | A final void will be done at 2 hours after the study drug discontinuation. The urine will be collected and volume recorded for each collection interval. |
| Whole body bio-impedance | | | | Prior to start of study drug infusion, at H4 (4 hours after the start of infusion and prior to furosemide bolus), at H8 (8 hours after the start of infusion and prior to study drug discontinuation), H10 (2 hours after the end of the infusion) in each treatment period. |
| Echocardiography | × | | × | Prior to start of study drug infusion, at H4 (4 hours after the start of infusion and prior to before furosemide bolus), at H5, H6, H8, and H10 (2 hours after the end of the infusion in each treatment period). |
| Lung ultrasound | × | | × | Prior to start of study drug infusion, at H4 (4 hours after the start of infusion and before furosemide bolus) and at H8 (end of infusion). |
| Clinical Drug Supplies | | | | |
| Randomize | × | | | Subjects will be randomized prior to start of infusion. Subjects will be randomized 1:1 to either BMS-986231 or Placebo in Period 1 and to either placebo or BMS-986231 in Period 2, such that within a sequence each patient will receive in random order one infusion of placebo. |
| Administration of Study Drug | × | | × | |
| Administration of furosemide bolus | × | | × | Furosemide bolus administration at H4 (4 hours after start of infusion of BMS-986231 or Placebo). |
| | | | - | |
| | | | _ | |





# **Appendix 3: Blood Sampling and Urine Collection Intervals for PK and Efficacy**

Blood sampling time points for furosemide, BMS-986231 (and its metabolites), Na and K are indicated as follows.

| Study Day of<br>Sample Collection<br>(of Each Period) | Event | Time (Relative To Start of Infusion<br>of BMS-986231)<br>Hour: Min | Blood Sample |
|---|---|---|---|
| 1 | Before start of infusion <sup>a</sup> | 00:00 | X |
| 1 | 2.0 hours <sup>a</sup> | 02:00 | X |
| 1 | 4.0 hours <sup>b</sup> | 04:00 | X |
| 1 | 5.0 hours | 05:00 | X |
| 1 | 6.0 hours | 06:00 | X |
| 1 | 8.0 hours (EOI) <sup>c</sup> | 08:00 | X |
| 1 | 10.0 | 10:00 | X |
| 1 | Dose lowered<br>due to safety<br>event | Misc. | X |

a this time-point is not applicable for furosemide analysis

EDSREP 009 T 01 G 

b just before furosemide bolus

<sup>&</sup>lt;sup>c</sup> EOI=End of Infusion, This sample should be taken immediately prior to stopping the infusion (preferably within 2 minutes prior to the end of infusion). If the end of infusion is delayed to beyond the nominal infusion duration, the collection of this sample should also be delayed accordingly.





Time points for urine collection intervals for Urine Output and Assessment of Furosemide, BMS-986231, K, Na, P, Bicarbonate, Creatinine, and Cl are as follows.

| Study Day of<br>Sample<br>Collection (of<br>Each Period) | Event | Time (Relative To<br>Start of Infusion of<br>BMS-986231)<br>Hour: Min | Urine Sample<br>Collection<br>Intervals <sup>a</sup> |
|---|---|---|---|
| 1 | Before start of infusion | 00:00 | X |
| 1 | 2.0 hours | 02:00 | 0-2 hours |
| 1 | 4.0 hours <sup>b</sup> | 04:00 | 2-4 hours |
| 1 | 5.0 hours | 05:00 | 4-5 hours |
| 1 | 6.0 hours | 06:00 | 5-6 hours |
| 1 | 7.0 hours | 07:00 | 6-7 hours |
| 1 | 8.0 hours (EOI) <sup>c</sup> | 08:00 | 7-8 hours |
| 1 | 10.0 hours | 10:00 | 8-10 hours |

a in the first 4 hours of the study drug infusion, and before furosemide bolus, urine collection will be done every 2 hours, thereafter the void will be hourly

EDSREP 009 T 01 G 

b just before furosemide bolus

EOI=End of Infusion, This sample should be taken immediately prior to stopping the infusion (preferably within 2 minutes prior to the end of infusion). If the end of infusion is delayed to beyond the nominal infusion duration, the collection of this sample should also be delayed accordingly.



Protocol: CV013-034 Version Date: 22-Jan-2020

| | ve | TSIOH Date: 22-Jan-2020 |
|---|----|-------------------------|
| | | # |
| _ | | |
| 1 | | |

EDSREP 009 T 01 G 


### Appendix 4: List of Tables, Figures, and Listings

| List of Tables and | Figures: | |
|---|---|---|
| Output | Title | Analysis Set |
| Section 14.1 – Disp | osition and Demographic Data | |
| Table 14.1.1 | Summary of Analysis Sets | All Subjects |
| Table 14.1.2 | Summary of Subject Disposition | All Subjects |
| Table 14.1.3.1 | Summary of Demographics | Randomized |
| Table 14.1.3.2 | Summary of Demographics | Per Protocol |
| Table 14.1.4 | Summary of Dosing | Safety |
| Section 14.2 – Efficacy Data | | |
| Table 14.2.1.1 | Summary of Urinary Output | Per Protocol |
| Figure 14.2.1.2 | Plot of Mean (+SD) Urinary Output over Time | Per Protocol |
| Figure 14.2.1.3.1 | Barchart of Mean Urinary Output over Time | Per Protocol |
| Figure 14.2.1.3.2 | Barchart of Individual Urinary Output over Time | Per Protocol |
| Table 14.2.1.4 | Statistical Analysis of the Volumes of Urinary Excretion | Per Protocol |
| Figure 14.2.1.5 | Plot of Paired Urinary Output by Treatment | Per Protocol |
| Figure 14.2.1.6 | Q-Q-Plot of Difference BMS-986231 – Placebo | Per Protocol |
| Table 14.2.2.1 | Summary of Fractional Excretion of FeNa and FeK | Per Protocol |
| Figure 14.2.2.2.1 | Barchart of Mean Fractional Excretion over Time | Per Protocol |
| Figure 14.2.2.2.2 | Barchart of Individual Fractional Excretion over Time | Per Protocol |
| Table 14.2.2.3 | Statistical Analysis of the Fractional Excretion | Per Protocol |
| Figure 14.2.2.4 | Plot of Paired Fractional Excretion | Per Protocol |
| Table 14.2.3.1 | Summary of Natriuresis | Randomized |
| Figure 14.2.3.2 | Plot of Paired Natriuresis | Randomized |
| Table 14.2.4.1 | Summary of Furosemide Concentration and Ratio of Urinary Sodium to Urinary Furosemide | Randomized |
| Figure 14.2.4.2 | Plot of Paired Furosemide Concentration and Ratio of Urinary Sodium to Urinary Furosemide | Randomized |
| Table 14.2.5 | Summary of eGFR and Creatinine Levels | Randomized |
| Table 14.2.6 | Summary of Renal and Urinary Biomarkers | Randomized |
| Table 14.2.7 | Summary of Body Weight | Randomized |
| Table 14.2.8 | Summary of Body Bio-Impedance | Randomized |
| Table 14.2.9 | Summary of Ultrasound Indices of Congestion | Randomized |
| Table 14.2.10 | Summary of Lung Ultrasound Indices of Pulmonary Congestion | Randomized |
| Table 14.2.11 | Summary of Pulmonary B-lines | Randomized |
| Section 14.2 – Phar | macokinetic Data | |
| Table 14.2.12.1 | Summary of Furosemide Plasma Concentrations | Randomized |
| Table 14.2.12.2 | Summary of Furosemide Urine Recovery by Interval | Randomized |

EDSREP 009 T 01 G 



Protocol: CV013-034 Version Date: 22-Jan-2020

| Table 14.2.12.3 | Summary of Furosemide Urine Recovery | Randomized |
|---|---|---|
| Table 14.2.12.4 | Summary of BMS-986231 and Metabolite Plasma Concentrations Randomized | |
| Table 14.2.12.5 | Summary of BMS-986231 and Metabolite Urine Recovery by Interval | Randomized |
| Section 14.3 – Safe | ty Data | |
| Table 14.3.1.1 | Summary of Adverse Events | Safety |
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term | Safety |
| Table 14.3.1.3 | Summary of Treatment Emergent Adverse Events by Relationship to Loestrin | Safety |
| Table 14.3.1.4 | Summary of Treatment Emergent Adverse Events by Relationship to BMS-986231 | Safety |
| Table 14.3.1.5 | Summary of Treatment Emergent Adverse Events by Severity | Safety |
| Table 14.3.2 | Listing of Deaths and Other Serious Adverse Events Enrolled | |
| Table 14.3.3 | Not part of TFL – Reserved for Narratives in CSR | |
| Table 14.3.4 | Listing of Abnormal Laboratory Values Enrolled | |
| Table 14.3.5 | Summary of Safety Laboratory Results Safety | |
| Table 14.3.6 | Summary of Vital Signs | Safety |
| Table 14.3.7 | Summary of 12-Lead Electrocardiogram Results | Safety |

| List of End of Text Listings: | |
|---|---|
| Output | Title |
| Section 16.2.1 – Dis | sposition |
| Listing 16.2.1.1 | Subject Disposition |
| Listing 16.2.1.2 | Eligibility Criteria |
| Section 16.2.2 – Pro | otocol Deviations |
| Listing 16.2.2 | Important Protocol Deviations |
| Section 16.2.3 – Ex | cluded Subjects |
| Listing 16.2.3 | Analysis Sets |
| Section 16.2.4 – De | mographics and Baseline Characteristics |
| Listing 16.2.4.1 | Subject Demographics |
| Listing 16.2.4.2 | Medical History |
| Listing 16.2.4.3 | Childbearing Potential |
| Listing 16.2.4.4 Prior and Concomitant Medications | |
| Section 16.2.5 - Compliance | |
| Listing 16.2.5.1 | Study Drug Administration – BMS986231 or Placebo |
| Listing 16.2.5.2 | Study Drug Administration – Furosemide |
| Section 16.2.6 – Re | sponse Data |
| Listing 16.2.6.1.1 | Urinary Output |

EDSREP 009 T 01 G 




|---|---|
| Listing 16.2.6.1.2 | Urinary Output - Differences |
| Listing 16.2.6.2.1 | Excretion of FeNa and FeK |
| Listing 16.2.6.2.2 | Fractional Excretion of FeNa and FeK - Differences |
| Listing 16.2.6.3.1 | Natriuresis |
| Listing 16.2.6.3.2 | Natriuresis - Differences |
| Listing 16.2.6.4.1 | Furosemide Concentration and Ratio of Urinary Sodium to Urinary Furosemide |
| Listing 16.2.6.4.2 | Furosemide Concentration and Ratio of Urinary Sodium to Urinary Furosemide - Differences |
| Listing 16.2.6.5.1 | eGFR and Creatinine Levels |
| Listing 16.2.6.5.2 | eGFR and Creatinine Levels – Differences |
| Listing 16.2.6.6.2 | Renal and Urinary Biomarkers – Differences |
| Listing 16.2.6.7.1 | Body Weight |
| Listing 16.2.6.7.2 | Body Weight – Differences |
| Listing 16.2.6.8.1 | Body Bio-Impedance |
| Listing 16.2.6.8.2 | Body Bio-Impedance – Differences |
| Listing 16.2.6.9.1 | Cardiac Ultrasound Indices of Congestion |
| Listing 16.2.6.9.2 | Cardiac Ultrasound Indices of Congestion – Differences |
| Listing 16.2.6.10.1 | Lung Ultrasound Indices of Pulmonary Congestion |
| Listing 16.2.6.10.2 | Lung Ultrasound Indices of Pulmonary Congestion – Differences |
| Listing 16.2.6.11.1 | Pulmonary B-lines |
| Listing 16.2.6.11.2 | Pulmonary B-lines – Differences |
| Section 16.2.7 – Pharmacokinetic Data | |
| Listing 16.2.7.1 | Listing of Furosemide Plasma Concentrations |
| Listing 16.2.7.2 | Listing of Furosemide Urine Concentrations |
| Listing 16.2.7.3 | Listing of Furosemide Urine Recovery |
| Listing 16.2.7.4 | Listing of BMS-986231 and Metabolite Plasma Concentrations |
| Listing 16.2.7.5 | Listing of BMS-986231 and Metabolite Urine Concentrations |
| Section 16.2.8 – Adverse Events Data | |
| Listing 16.2.8.1 | Adverse Events |
| Listing 16.2.8.2 | Adverse Events Resulting in Study Drug Discontinuation |
| Section 16.2.9 – La | boratory Data |
| Listing 16.2.9.1 | Clinical Laboratory Results – Chemistry |
| Listing 16.2.9.2 | Clinical Laboratory Results – Hematology |
| Listing 16.2.9.3 | Clinical Laboratory Results – Pregnancy Test |
| Section 16.2.10 On | ward – Other Safety Data |
| Listing 16.2.10.1 | Vital Signs |
| Listing 16.2.10.2 | Hypotension |

EDSREP 009 T 01 G 




| Listing 16.2.11 | 12-Lead Electrocardiogram Results |
|-----------------|-----------------------------------|
| Listing 16.2.12 | Physical Examinations |

| Other Appendix O | utputs: |
|-------------------|------------------------|
| Output | Title |
| Appendix 16.1.9.2 | Statistical Appendices |

EDSREP 009 T 01 G 




### **Appendix 6: Shells for Tables, Figures and Listings**

Shells are provided in a separate document.

EDSREP 009 T 01 G 




### **18.0 Document History**

| Version Date | Modified/Reviewed By | Brief Summary of Changes |
|---|---|---|
| 13-Dec-2019 | | Created from EDSREP 009 T 01 G including agreements for the PRA/ BMS Phase I work. |
| 20-Dec-2019 | | Implemented comments from internal review |
| 22-Jan-2020 | | Implemented comments from internal and sponsor review |

EDSREP 009 T 01 G 